CLINICAL TRIAL: NCT03650959
Title: Optimizing Resource Utilization During Proficiency-Based Training of Suturing Skills to Medical Students: a Randomized Controlled Trial of Faculty-Led, Peer Tutor-Led, and Computer Augmented Methods of Teaching
Brief Title: Optimizing Resource Utilization During Proficiency-based Training of Suturing Skills to Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Boris Zevin, Assistant Professor & Medical Education Scholar, Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SURG-422-18
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2018-08

CONDITIONS: Education, Medical; Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Faculty-led (Experimental)
  Interventions: Other: Method of learning simple interrupted sutures with instrument tie
- Peer tutor-led (Experimental)
  Interventions: Other: Method of learning simple interrupted sutures with instrument tie
- Computer augmented self-directed learning (Experimental)
  Interventions: Other: Method of learning simple interrupted sutures with instrument tie

INTERVENTIONS:
Other: Method of learning simple interrupted sutures with instrument tie — Students will train to proficiency (defined by hand motion analysis) on simple interrupted sutures with an instrument tie via one of three different methods: faculty-led, peer tutor-led, or computer augmented self-directed learning.

SUMMARY:
Evidence favours teaching procedural skills to medical students using a proficiency-based rather than time-based approach. Basic suturing skills can be taught through faculty-led, peer tutor-led, and computer augmented approaches. One method has yet to be identified as superior in terms of educational outcomes, resource utilization, and participant perspectives.

Pre-clerkship medical students were randomized to: faculty, peer tutor, or computer augmented learning. Participants practiced suturing through their randomized method until they reached targeted proficiency defined using hand motion analysis (HMA). Proficiency was defined as a score of the average plus a standard deviation of five surgeons' HMA for two of three consecutive sutures using appropriate technique.

The primary outcome was the number of stitches placed to achieve proficiency. The secondary outcomes were the number of sutures used, time, and costs incurred. Learning curves were constructed. Participants' perceptions were assessed using a follow-up survey.

ELIGIBILITY:
Inclusion Criteria:

* Second year, pre-clerkship medical students

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-06-16 (Actual); Study Completion 2019-06-16 (Actual)

PRIMARY OUTCOMES:
Number of stitched laid to reach proficiency | Five days

SECONDARY OUTCOMES:
Number of sutures used to reach proficiency | Five days
Minutes to reach proficiency | Five days
Individual costs to reach proficiency | Five days

OTHER OUTCOMES:
Learning curves | Five days
Student preferences | Five days

CONTACTS AND LOCATIONS:
Locations (1):
- Queen's Unviersity, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No